CLINICAL TRIAL: NCT02873234
Title: A Multicentre Prospective Cohort Study of Traditional Chinese Medicine Treating Depression With The Use of Cloud Data
Brief Title: A Study of Chinese Medicine Treating Depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Third Affiliated Hospital of Beijing University of Chinese Medicine (Other)
Collaborators: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other); Beijing HuiLongGuan Hospital (Other); The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); First Affiliated Hospital of Heilongjiang Chinese Medicine University (Other); The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other); Shandong University of Traditional Chinese Medicine (Other); Capital Medical University (Other); Xiamen Hospital of Traditional Chinese Medicine (Other); Wu Xi Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Qisheng Tang, MD, PHD, The Third Affiliated Hospital of Beijing University of Chinese Medicine
Other Study IDs: 201507001-12
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Depression
Keywords: Telemedicine; Chinese Medicine syndrome differentiation; Long-term study; Relapse rate; Suicide rate; Antidepressants
MeSH Terms: conditions — Depression | interventions — Medicine, Chinese Traditional; Antidepressive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Traditional Chinese Medicine: Including Zishui Qinggan Yin,Xiaoyao San, Longdan Xiegan Tang, Guipi Decoction, Ningshen Dingzhi Wan, HuangLian-EJiao decoction and Jiaotai Wan.
  Interventions: Drug: Traditional Chinese Medicine
- TCM plus antidepressants: This is a integrative therapy that refers to a new treating system including TCM and antidepressants.
  Interventions: Drug: Traditional Chinese Medicine; Drug: Antidepressants
- Antidepressants: Antidepressants include Selective serotonin reuptake inhibitors (SSRIs), Norepinephrine-reuptake inhibitors and other antidepressants, such as Paroxetine, Citalopram, Venlafaxine, Sertraline, Trazodone, Maprotiline and so on.
  Interventions: Drug: Antidepressants

INTERVENTIONS:
Drug: Traditional Chinese Medicine — Participants are treated with TCM twice per day according to syndrome differentiation. For example, the syndrome of one participant with depression is kidney deficiency. He will take Zishui Qinggan Yin twice per day before the breakfast and dinner.
  Other Names: Chinese Medicine, Chinese Herb Medicine
  Groups: TCM plus antidepressants; Traditional Chinese Medicine
Drug: Antidepressants — Participants are treated with different antidepressants. The dosage, frequency and duration are determined according to guideline.
  Groups: Antidepressants; TCM plus antidepressants

SUMMARY:
Chinese Medicine syndrome differentiation has been a prevalent therapy in China for thousands of years. It is based on patients' symptoms, pulse, tongue and coating on the tongue. Therefore, the syndrome of patients and corresponding Traditional Chinese Medicine (TCM) may vary.

This multicenter prospective cohort studies the efficiency and safety of TCM compared with antidepressants. A total number of 4600 cases with primary depression are expected to be collected and divided into 3 cohorts based on the patients' requirement and choices. Patients in one group will receive TCM, and patients in the other two groups will respectively receive antidepressants only and integrated treatment of TCM and antidepressants. This study has 2 phases: treating period and the follow-up.

The main purpose of this long-term study is to evaluate the efficiency of TCM compared with antidepressants in reducing relapse and suicide rate, changing lifestyle, improving patient compliance as well as the safety.

DETAILED DESCRIPTION:
This multicenter prospective cohort uses a modern technique. With its help participants can assess themselves at any time and doctors can supervise patients in case of some adverse events or intervene when patients commit suicide.

The main purpose of this study is to observe the differences between cohorts. However, the intra-group differences are also needed to be evaluated, as the therapies of different participants are various. Therefore, the number of participants treated with each therapy and the time of recovery need to be counted and analyzed. This is a long-term and natural study that participants lost, drug withdrawal and changes in participants'choices of the therapy cannot be avoided. So the reason and number of the previous conditions need to be observed. The safety of TCM and antidepressants is also a considerable outcome which will be evaluated by laboratory examination, Treatment Emergent Symptom Scale (TESS) and the number of participants with adverse events.

Some of the outcomes are measured by questionnaires which can be divided into two parts. One is self-rated assessments including Self-rating Depression Scale (SDS) and Self-reporting Inventory (SCL-90). The other one is evaluated by doctors, such as Hamilton Depression Rating Scale of 24 items (HAMD), Montgomery-Asberg Depression Rating Scale (MADRS), Social Disability Screening Schedule (SDSS), Mini-mental State Examination (MMSE), Montreal Cognitive Assessment (MoCA)and Traditional Chinese Medicine syndrome score.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria can be included in this study:

* Clinical diagnosis of depression
* The scores of Hamilton Depression scale ( HAMD )≥18
* With stable vital signs, conscious mind and acceptable communication ability
* Can use the mobile phone to do self-evaluation
* Male or female patients between 18 and 65 years old
* Signing the informed consent and agreeing to participate in this study

Exclusion Criteria:

Subjects meeting anyone of the following criteria will be excluded from this study:

* Depression caused by other diseases
* Unstable vital signs
* Severe aphasia and agnosia causing disability to communicate
* Alcoholism and other substance dependence
* Diagnosis of other mental disorders except depression
* Serious hepatic or renal insufficiency
* Pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Depressive subjects with proven primary depression will be asked to participate in this study.
Sampling Method: Probability Sample
Enrollment: 4600 (Estimated)
Dates: Start 2016-06; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Relapse rate | 2 years
  It is the percentage of the relapse of depression including the total number of relapse cases.
Suicide rate | 2 years
  The suicide rate includes the percentage of the cases committing suicide and the successful cases.

SECONDARY OUTCOMES:
Self-rating Depression Scale (SDS) | 2 years
  Differences between groups are evaluated by the change of total scores from the study starting to every 2 weeks at least during 2 years. It is assessed by patients using a mobile phone APP.
Self-reporting Inventory (SCL-90) | 2 years
  Differences between groups are evaluated by the change of total scores from the study starting to every 2 weeks at least during 2 years. It is assessed by patients using a mobile phone APP.
Hamilton Depression Rating Scale of 24 items (HAMD) | before recruiting
  Differences between groups are evaluated by change of total scores from the study intake to every 3 months in 2 years.
Social Disability Screening Schedule (SDSS) | 2 years
  Differences between groups are evaluated by change of total scores from the study intake to every 3 months in 2 years.
Traditional Chinese Medicine syndrome score | 2 years
  Before the study, all investigators took standardized training and conformance testing. Syndrome differentiation and syndrome scores were took by 2 investigators together, and the results needed to obtain their consent.
Recovery Rate | 2 years
  The differences between groups are evaluated by the number and rate of recovery cases from the study intake to every 3 months in 2 years.
Montgomery-Asberg Depression Rating Scale (MADRS) | 2 years
  Differences between groups are evaluated by change of total scores from the study intake to every 3 months in 2 years.
Mini-mental State Examination (MMSE) | 2 years
  Differences between groups are evaluated by change of total scores from the study intake to every 3 months in 2 years.
Montreal Cognitive Assessment Scale (MoCA) | 2 years
  Differences between groups are evaluated by change of total scores from the study intake to every 3 months in 2 years.
The time of relapse | 2 years
The time of committing suicide | 2 years
  It refers to the time of committing suicide and the time of success.

OTHER OUTCOMES:
Laboratory examination | 2 years
  Blood RT, Hepatic function and Renal function
Treatment Emergent Symptom Scale (TESS) | 2 years
  TESS documents the presence of common side effects. Low scores or decrease in scores represent less side effects and high scores or increase in scores represent more side effects.
Number of participants with adverse events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Qisheng Tang, MD, PHD, Study Director — The Third Affiliated Hospital of Beijing University of Chinese Medicine
Locations (1):
- The Third Affiliated Hospital of Beijing University of Chinese Medicine, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No